CLINICAL TRIAL: NCT05648422
Title: Effect of the Nutritional Support System (NSS) on Neuromotor Alterations in Patients With Cerebral Palsy
Brief Title: Effect of the Nutritional Support System on Neuromotor Alterations in Patients With Cerebral Palsy
Acronym: NSS-PC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Anahuac University (Other)
Responsible Party: Principal Investigator, Fernando Leal-Martinez, Principal investigator, Anahuac University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: 202082
Record Dates: First submitted 2022-02-15; First posted 2022-12-13 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy; Spastic; Malnutrition
Keywords: Cerebral Palsy; Nutritional Support; NSS; Probiotics; Diet; Neurogenesis; Neuroplasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity; Malnutrition | interventions — Probiotics; nitazoxanide; World Health Organization

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial with blinding.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The outcomes assessors and care providers had no access to any information about the treatment administered to each child, which ensured compliance with the blinded portion of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- FG (FOLLOW GROUP) (No Intervention): FG receive: Conventional diet (WHO).
- CG (CONTROL GROUP) (Experimental): CG receive: Conventional diet (WHO), deworming (nitazoxanide at a dosage of 7.5 mg / kg every 12 hours for 3 days), and probiotics (Saccharomyces Boulardii, 200 mg every 12 hours for 6 days at week 1, 5 and 9).
  Interventions: Dietary Supplement: Probiotics; Drug: Deworming; Other: Conventional diet (WHO)
- IG (INTERVENTION GROUP) (Experimental): IG receive: Deworming (nitazoxanide at a dosage of 7.5 mg / kg every 12 hours for 3 days), probiotics (Saccharomyces Boulardii, 200 mg every 12 hours for 6 days at week 1, 5 and 9), specific diet, and NSS envelope (glutamine, arginine, folic acid, PUFA-n3, vegetal protein, nicotinic acid, cobalamin, thiamine, pyridoxine, magnesium, zinc, selenium, cholecalciferol, resveratrol, ascorbic acid, Spirulina Máxima, and inuline) every 12 hours for 12 weeks.
  Interventions: Dietary Supplement: Probiotics; Dietary Supplement: NSS Nutritional Support System; Drug: Deworming; Other: Specific diet

INTERVENTIONS:
Dietary Supplement: Probiotics — Saccharomyces Boulardii 200 mg every 12 hours for 6 days at week 1, 5 and 9
  Other Names: Probiotics (Saccharomyces Boulardii)
  Arms: CG (CONTROL GROUP); IG (INTERVENTION GROUP)
Dietary Supplement: NSS Nutritional Support System — Nutritional Support System consists in NSS envelope (glutamine, arginine, folic acid, PUFA-n3, vegetal protein, nicotinic acid, cobalamin, thiamine, pyridoxine, magnesium, zinc, selenium, cholecalciferol, resveratrol, ascorbic acid, Spirulina Máxima, glycine, tryptophan, and inuline) every 12 hours for 12 weeks.
  Other Names: NSS
  Arms: IG (INTERVENTION GROUP)
Drug: Deworming — nitazoxanide at a dosage of 7.5 mg / kg every 12 hours for 3 days
  Other Names: Nitazoxanide
  Arms: CG (CONTROL GROUP); IG (INTERVENTION GROUP)
Other: Specific diet — This diet focuses on meeting caloric needs according to age, weight, height, and stress factor dividing total caloric value in 50% carbohydrates, 30% lipids, and 20% proteins. It consists of smoothies at breakfast and dinner, high consumption of fish, five meals during the day, 70% of meals eaten during the day will consist on vegetables, fruits, roots, cereals, and legumes. Red meat, gluten, lactose, junk food, sugar, salt, fast food free.
  Arms: IG (INTERVENTION GROUP)
Other: Conventional diet (WHO) — This diet focuses on meeting caloric needs according to age, weight, height, and stress factor dividing total caloric value in 50% carbohydrates, 30% lipids, and 20% proteins. It consists of general nutricional recommendations.
  Arms: CG (CONTROL GROUP)

SUMMARY:
Study to determine the impact of a nutritional support system (NSS) on neuromotor alterations in patients with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a group of motor disorders of the brain and can be accompanied by alterations in sensation, perception, cognition, communication and behavior, epilepsy and secondary musculoskeletal disorders. These disorders decrease daily functional performance in the areas of mobility, cognition and self-care, resulting in the need for a primary caregiver and increased health care costs. Rehabilitative treatment to increase functional independence is taken from the point of view of motor function (physiotherapy), however, no emphasis is placed on nutritional treatment aimed at alterations in mobility, cognition and self-care; currently it has been observed that eating disorders alter neuromuscular function directly or indirectly, therefore many patients do not respond adequately to treatment due to deterioration in secondary nutritional status. Dietary deficiency in patients with ICH is the result of the lack of an essential nutrient in the diet, each of these nutrients has a functional dynamic in the different stages, so that if one of them is missing or deficient, a functional or organic alteration, a biochemical variation or a disorder in body mass will occur. The World Health Organization (WHO) only considers energy, protein and fat requirements according to the age of the child. The NSS (Nutritional Support System) consisting of specific diet, supplementation (glutamine, arginine, folic acid, PUFA-n3, vegetal protein, nicotinic acid, cobalamin, thiamine, pyridoxine, magnesium, zinc, selenium, cholecalciferol, resveratrol, ascorbic acid, Spirulina Máxima, and inuline) and probiotics, have individually demonstrated effects such as neuronal regeneration, neuroprotective effect, reduction of oxidative stress.

A randomized, blinded, clinical trial will be conducted in children aged 4 to 11 years with CP functional level III of the Gross Motor Function Classification System (GMFCS), without impaired cognitive status and unable to walk on their own. They are randomly assigned to three groups: 1) follow-up group (GS) to which conventional diet (WHO) be applied; 2) control group 2 (GC) to which conventional diet (WHO), deworming and probiotics will be applied 3) intervention group (GI) deworming, probiotics, NSS supplements and specific diet will be applied, they will be followed up for three months; They will be evaluated at baseline, week 7 and week 13 with Gross Motor Function Measure 66 (GMFM-66) and MACS; at baseline and week 13 with kinetics and kinematic analysis, and electromyography (EMG). Statistical analysis: For the intragroup inferential statistical analysis, 2-way ANOVA will be used if the distribution is normal, otherwise FRIEDMAN will be used, in both cases post hoc tests will be applied; for the intergroup analysis, 1-way ANOVA will be used if the distribution is normal, otherwise KRUSKAL WALLIS will be used, in both cases post hoc tests will be applied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GMFCS III classification.
* Patients with spastic CP.
* Both sexes age 4 to 11 years.
* Primary caregiver engaged (full presence).
* Able to follow instructions.
* Tolerant to oral feeding.
* Parents or guardians to sign informed consent letter.
* Children, if able to write, sign the letter of assent.

Exclusion Criteria:

* Have received antibiotics 15 days prior to treatment.
* Having received botulinum toxin therapy in the last six months. Consumption of muscle relaxants in the last three months.
* Patient with any type of surgery in a period of less than 6 months.
* Presence of any other catabolic disease, which further increases their risk of malnutrition (renal, cardiovascular, pulmonary, hepatic, immunological).
* Intolerance to oral feeding.
* Lack of stimulation at home.
* Moderate to severe gastroesophageal reflux.
* Able to walk without support.

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
CHANGE FROM BASELINE GROSS MOTOR FUNCTION MEASURE 66 AT 7 WEEKS | Baseline period, and week 7
  It measures five mobility ability areas, known as dimensions: lying, sitting, crawling and kneeling, standing, and walking, running and jumping.
  The main criterion is that the difference between each level is significant for daily living and these are based on functional limitations, support from gait aids such as crutches, canes, walkers or wheeled mobility.
  It is intended to indicate at what level the child/youth's gross motor functioning abilities and limitations are at.
CHANGE FROM BASELINE GROSS MOTOR FUNCTION MEASURE 66 AT 13 WEEKS | Baseline period, and week 13
  It measures five mobility ability areas, known as dimensions: lying, sitting, crawling and kneeling, standing, and walking, running and jumping.
  The main criterion is that the difference between each level is significant for daily living and these are based on functional limitations, support from gait aids such as crutches, canes, walkers or wheeled mobility.
  It is intended to indicate at what level the child/youth's gross motor functioning abilities and limitations are at.
CHANGE FROM BASELINE MANUAL ABILITY CLASSIFICATION SYSTEM AT 7 WEEKS | Baseline period, week 7
  The Manual Ability Classification System (MACS) is a functional description and is also used to complement the child's diagnostic assessment giving a classification based on fine motor skills.
  The MACS results are based on the child's performance in daily life, it does not take into account the differences between the function of the two hands; rather, it looks at how children handle age-appropriate objects and the need and extent of support or adaptations.
CHANGE FROM BASELINE MANUAL ABILITY CLASSIFICATION SYSTEM 13 WEEKS | Baseline period, week 13
  The Manual Ability Classification System (MACS) is a functional description and is also used to complement the child's diagnostic assessment giving a classification based on fine motor skills.
  The MACS results are based on the child's performance in daily life, it does not take into account the differences between the function of the two hands; rather, it looks at how children handle age-appropriate objects and the need and extent of support or adaptations.
CHANGE FROM BASELINE MUSCLE ELECTRIC ACTIVITY AT 13 WEEKS | Baseline and week 13
  This study will measure the average behavior of a muscle or muscle group. It will give information on spasticity, coactivation of synergic and antagonic muscles, and maximum voluntary contraction.
  The changes at muscle electric activity will be evaluated by applying electromyography (EMG) studies at baseline and at week 13.
CHANGE FROM BASELINE GAIT ANALYSIS AT 13 WEEKS | Baseline and week 13
  This will provide objective and quantitative measures useful to assess gross motor skills with spatiotemporal, kinetics and kinematics data.
  In each gait cycle it will measure walking speed, cadence, stride and step length and support, and joint angles.
  The progression of the patient from the baseline period compared to week 13 will be evaluated with 3D motion capture systems.
CHANGE FROM BASELINE CRAWLING ANALYSIS AT 13 WEEKS | Baseline and week 13
  This will provide objective and quantitative measures useful to assess gross motor skills with spatiotemporal, kinetics and kinematics data.
  In each crawling analysis, speed, inter limb coordination and joint angles will be measured with 3D motion capture systems.

SECONDARY OUTCOMES:
CHANGE FROM BASELINE MIDARM MUSCLE AREA AT 7 WEEKS | Baseline and week 7
  Midarm muscle area (MMA) will be calculated using the equation: [MCA - (π (TSF))^2]/4π) Mid upper arm circumference (MCA) will be measured in centimeters and the tricipital skinfold (TSF) will be measured using Harpenden skin fold caliper giving the measurements in millimeters.
CHANGE FROM BASELINE MIDARM MUSCLE AREA AT 13 WEEKS | Baseline and week 13
  Midarm muscle area (MMA) will be calculated using the equation: [MCA - (π (TSF))^2]/4π) Mid upper arm circumference (MCA) will be measured in centimeters and the tricipital skinfold (TSF) will be measured using Harpenden skin fold caliper giving the measurements in millimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Leal, PhD, Study Director — Anahuac University
Locations (1):
- Apac I.A.P. (Association For People With Cerebral Palsy), México, Mexico

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers whose proposed use of the data has been approved by an independent review committee identified for this purpose.
  Proposals should be directed to ferman5@hotmail.com.

REFERENCES:
- [Background] Trotta T, Porro C, Cianciulli A, Panaro MA. Beneficial Effects of Spirulina Consumption on Brain Health. Nutrients. 2022 Feb 5;14(3):676. doi: 10.3390/nu14030676. PMID 35277035
- [Background] Schweizer U, Fabiano M. Selenoproteins in brain development and function. Free Radic Biol Med. 2022 Sep;190:105-115. doi: 10.1016/j.freeradbiomed.2022.07.022. Epub 2022 Aug 10. PMID 35961466
- [Background] Roy Sarkar S, Mitra Mazumder P, Chatterjee K, Sarkar A, Adhikary M, Mukhopadhyay K, Banerjee S. Saccharomyces boulardii ameliorates gut dysbiosis associated cognitive decline. Physiol Behav. 2021 Jul 1;236:113411. doi: 10.1016/j.physbeh.2021.113411. Epub 2021 Mar 31. PMID 33811908
- [Background] Visco DB, Toscano AE, Juarez PAR, Gouveia HJCB, Guzman-Quevedo O, Torner L, Manhaes-de-Castro R. A systematic review of neurogenesis in animal models of early brain damage: Implications for cerebral palsy. Exp Neurol. 2021 Jun;340:113643. doi: 10.1016/j.expneurol.2021.113643. Epub 2021 Feb 23. PMID 33631199
- [Background] Rubin DI. Needle Electromyography Waveforms During Needle Electromyography. Neurol Clin. 2021 Nov;39(4):919-938. doi: 10.1016/j.ncl.2021.06.003. Epub 2021 Aug 31. PMID 34602219
- [Background] Le Roy C, Barja S, Sepulveda C, Guzman ML, Olivarez M, Figueroa MJ, Alvarez M. Vitamin D and iron deficiencies in children and adolescents with cerebral palsy. Neurologia (Engl Ed). 2021 Mar;36(2):112-118. doi: 10.1016/j.nrl.2017.11.005. Epub 2018 Jan 17. English, Spanish. PMID 29342407
- [Background] Tinkov AA, Skalnaya MG, Skalny AV. Serum trace element and amino acid profile in children with cerebral palsy. J Trace Elem Med Biol. 2021 Mar;64:126685. doi: 10.1016/j.jtemb.2020.126685. Epub 2020 Nov 12. PMID 33249374
- [Background] Huff TC, Sant DW, Camarena V, Van Booven D, Andrade NS, Mustafi S, Monje PV, Wang G. Vitamin C regulates Schwann cell myelination by promoting DNA demethylation of pro-myelinating genes. J Neurochem. 2021 Jun;157(6):1759-1773. doi: 10.1111/jnc.15015. Epub 2020 Apr 14. PMID 32219848
- [Background] Sorrenti V, Castagna DA, Fortinguerra S, Buriani A, Scapagnini G, Willcox DC. Spirulina Microalgae and Brain Health: A Scoping Review of Experimental and Clinical Evidence. Mar Drugs. 2021 May 22;19(6):293. doi: 10.3390/md19060293. PMID 34067317
- [Background] Eyles DW. Vitamin D: Brain and Behavior. JBMR Plus. 2020 Oct 18;5(1):e10419. doi: 10.1002/jbm4.10419. eCollection 2021 Jan. PMID 33553986
- [Background] Kazmierczak-Siedlecka K, Ruszkowski J, Fic M, Folwarski M, Makarewicz W. Saccharomyces boulardii CNCM I-745: A Non-bacterial Microorganism Used as Probiotic Agent in Supporting Treatment of Selected Diseases. Curr Microbiol. 2020 Sep;77(9):1987-1996. doi: 10.1007/s00284-020-02053-9. Epub 2020 May 29. PMID 32472262
- [Background] Sainz-Pelayo MP, Albu S, Murillo N, Benito-Penalva J. [Spasticity in neurological pathologies. An update on the pathophysiological mechanisms, advances in diagnosis and treatment]. Rev Neurol. 2020 Jun 16;70(12):453-460. doi: 10.33588/rn.7012.2019474. Spanish. PMID 32500524
- [Background] Sadowska M, Sarecka-Hujar B, Kopyta I. Cerebral Palsy: Current Opinions on Definition, Epidemiology, Risk Factors, Classification and Treatment Options. Neuropsychiatr Dis Treat. 2020 Jun 12;16:1505-1518. doi: 10.2147/NDT.S235165. eCollection 2020. PMID 32606703
- [Background] Vitrikas K, Dalton H, Breish D. Cerebral Palsy: An Overview. Am Fam Physician. 2020 Feb 15;101(4):213-220. PMID 32053326
- [Background] Leal-Martinez F, Franco D, Pena-Ruiz A, Castro-Silva F, Escudero-Espinosa AA, Rolon-Lacarrier OG, Lopez-Alarcon M, De Leon X, Linares-Eslava M, Ibarra A. Effect of a Nutritional Support System (Diet and Supplements) for Improving Gross Motor Function in Cerebral Palsy: An Exploratory Randomized Controlled Clinical Trial. Foods. 2020 Oct 13;9(10):1449. doi: 10.3390/foods9101449. PMID 33066040
- [Background] Choi S, Hong DK, Choi BY, Suh SW. Zinc in the Brain: Friend or Foe? Int J Mol Sci. 2020 Nov 25;21(23):8941. doi: 10.3390/ijms21238941. PMID 33255662
- [Background] Santos HO, Teixeira FJ, Schoenfeld BJ. Dietary vs. pharmacological doses of zinc: A clinical review. Clin Nutr. 2020 May;39(5):1345-1353. doi: 10.1016/j.clnu.2019.06.024. Epub 2019 Jul 4. PMID 31303527
- [Background] Hariharan S, Dharmaraj S. Selenium and selenoproteins: it's role in regulation of inflammation. Inflammopharmacology. 2020 Jun;28(3):667-695. doi: 10.1007/s10787-020-00690-x. Epub 2020 Mar 6. PMID 32144521
- [Background] Calderon-Ospina CA, Nava-Mesa MO. B Vitamins in the nervous system: Current knowledge of the biochemical modes of action and synergies of thiamine, pyridoxine, and cobalamin. CNS Neurosci Ther. 2020 Jan;26(1):5-13. doi: 10.1111/cns.13207. Epub 2019 Sep 6. PMID 31490017
- [Background] Michielsen M, Vaughan-Graham J, Holland A, Magri A, Suzuki M. The Bobath concept - a model to illustrate clinical practice. Disabil Rehabil. 2019 Aug;41(17):2080-2092. doi: 10.1080/09638288.2017.1417496. Epub 2017 Dec 17. PMID 29250987
- [Background] Vinals-Labanino CP, Velazquez-Bustamante AE, Vargas-Santiago SI, Arenas-Sordo ML. Usefulness of Cerebral Palsy Curves in Mexican Patients: A Cross-Sectional Study. J Child Neurol. 2019 May;34(6):332-338. doi: 10.1177/0883073819830560. Epub 2019 Mar 11. PMID 30854918
- [Background] Fragale N, Navarre N, Rogers J. General Nutrition for Children with Cerebral Palsy. In: Miller F, Bachrach S, Lennon N, O'Neil M, editors. Cerebral Palsy Cham: Springer International Publishing; 2019. p. 1-10.
- [Background] Steele KM, Munger ME, Peters KM, Shuman BR, Schwartz MH. Repeatability of electromyography recordings and muscle synergies during gait among children with cerebral palsy. Gait Posture. 2019 Jan;67:290-295. doi: 10.1016/j.gaitpost.2018.10.009. Epub 2018 Oct 22. PMID 30396059
- [Background] Picon-Pages P, Garcia-Buendia J, Munoz FJ. Functions and dysfunctions of nitric oxide in brain. Biochim Biophys Acta Mol Basis Dis. 2019 Aug 1;1865(8):1949-1967. doi: 10.1016/j.bbadis.2018.11.007. Epub 2018 Nov 27. PMID 30500433
- [Background] Kaur H, Bose C, Mande SS. Tryptophan Metabolism by Gut Microbiome and Gut-Brain-Axis: An in silico Analysis. Front Neurosci. 2019 Dec 18;13:1365. doi: 10.3389/fnins.2019.01365. eCollection 2019. PMID 31920519
- [Background] Lu J, Claud EC. Connection between gut microbiome and brain development in preterm infants. Dev Psychobiol. 2019 Jul;61(5):739-751. doi: 10.1002/dev.21806. Epub 2018 Nov 20. PMID 30460694
- [Background] Panti-May JA, Zonta ML, Cociancic P, Barrientos-Medina RC, Machain-Williams C, Robles MR, Hernandez-Betancourt SF. Occurrence of intestinal parasites in Mayan children from Yucatan, Mexico. Acta Trop. 2019 Jul;195:58-61. doi: 10.1016/j.actatropica.2019.04.023. Epub 2019 Apr 22. PMID 31022382
- [Background] Bivona G, Gambino CM, Iacolino G, Ciaccio M. Vitamin D and the nervous system. Neurol Res. 2019 Sep;41(9):827-835. doi: 10.1080/01616412.2019.1622872. Epub 2019 May 30. PMID 31142227
- [Background] Gasperi V, Sibilano M, Savini I, Catani MV. Niacin in the Central Nervous System: An Update of Biological Aspects and Clinical Applications. Int J Mol Sci. 2019 Feb 23;20(4):974. doi: 10.3390/ijms20040974. PMID 30813414
- [Background] Ballaz SJ, Rebec GV. Neurobiology of vitamin C: Expanding the focus from antioxidant to endogenous neuromodulator. Pharmacol Res. 2019 Aug;146:104321. doi: 10.1016/j.phrs.2019.104321. Epub 2019 Jun 20. PMID 31229562
- [Background] Heshmati J, Morvaridzadeh M, Maroufizadeh S, Akbari A, Yavari M, Amirinejad A, Maleki-Hajiagha A, Sepidarkish M. Omega-3 fatty acids supplementation and oxidative stress parameters: A systematic review and meta-analysis of clinical trials. Pharmacol Res. 2019 Nov;149:104462. doi: 10.1016/j.phrs.2019.104462. Epub 2019 Sep 26. PMID 31563611
- [Background] Tamtaji OR, Heidari-Soureshjani R, Mirhosseini N, Kouchaki E, Bahmani F, Aghadavod E, Tajabadi-Ebrahimi M, Asemi Z. Probiotic and selenium co-supplementation, and the effects on clinical, metabolic and genetic status in Alzheimer's disease: A randomized, double-blind, controlled trial. Clin Nutr. 2019 Dec;38(6):2569-2575. doi: 10.1016/j.clnu.2018.11.034. Epub 2018 Dec 10. PMID 30642737
- [Background] Sharma SK, Bansal MP, Sandhir R. Altered dietary selenium influences brain iron content and behavioural outcomes. Behav Brain Res. 2019 Oct 17;372:112011. doi: 10.1016/j.bbr.2019.112011. Epub 2019 Jun 15. PMID 31212061
- [Background] Gao Z, Chen L, Xiong Q, Xiao N, Jiang W, Liu Y, Wu X, Hou W. Degraded Synergistic Recruitment of sEMG Oscillations for Cerebral Palsy Infants Crawling. Front Neurol. 2018 Sep 18;9:760. doi: 10.3389/fneur.2018.00760. eCollection 2018. PMID 30279674
- [Background] Caramico-Favero DCO, Guedes ZCF, Morais MB. FOOD INTAKE, NUTRITIONAL STATUS AND GASTROINTESTINAL SYMPTOMS IN CHILDREN WITH CEREBRAL PALSY. Arq Gastroenterol. 2018 Oct-Dec;55(4):352-357. doi: 10.1590/S0004-2803.201800000-78. PMID 30785518
- [Background] Guo YE, Suo N, Cui X, Yuan Q, Xie X. Vitamin C promotes oligodendrocytes generation and remyelination. Glia. 2018 Jul;66(7):1302-1316. doi: 10.1002/glia.23306. Epub 2018 Feb 9. PMID 29423921
- [Background] Garcia-Sanchez SF, Gomez-Galindo MT, Guzman-Pantoja JE. [Botulinum toxin A and physical therapy in gait in cerebral palsy]. Rev Med Inst Mex Seguro Soc. 2017 Jan-Feb;55(1):18-24. Spanish. PMID 28092243
- [Background] Westfall S, Lomis N, Kahouli I, Dia SY, Singh SP, Prakash S. Microbiome, probiotics and neurodegenerative diseases: deciphering the gut brain axis. Cell Mol Life Sci. 2017 Oct;74(20):3769-3787. doi: 10.1007/s00018-017-2550-9. Epub 2017 Jun 22. PMID 28643167